CLINICAL TRIAL: NCT05807672
Title: MARF-E- Magnetic Resonance Fingerprinting in the Imaging of Endometrial Cancer
Brief Title: Magnetic Resonance Fingerprinting in the Imaging of Endometrial Cancer
Acronym: MARF-E
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 4690
Record Dates: First submitted 2023-03-06; First posted 2023-04-11 (Actual); Last update posted 2023-04-11 (Actual); Status verified 2023-03

CONDITIONS: Endometrial Cancer
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In this context, the aim of this study is to investigate the role of MRF in endometrial cancer. Several applications are possible. Firstly, T1-, T2- and DWI-mappings can be associated to molecular risk group classification, in order to stratify patients' risk without recurring to surgery. MRF parameters can be also correlated to prognosis, both in terms of disease-free survival (DFS) and overall survival (OS).

ELIGIBILITY:
Inclusion Criteria:

* Patients with biopsy-proven endometrial cancer;
* Women aged > 18 years old;
* Signed Informed consent.

Exclusion Criteria:

* Previous history of neoplasm;
* Concurrent malignancies at other sites.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients that undergo to clinics/hospitalization examination at Fondazione Policlinico Universitario "A. Gemelli" IRCCS for endometrial cancers will be candidate to partecipate to this study, according to exclusion and inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2022-04-23 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Association between T1-, T2- and diffusion-mappings and risk group classification | 3 months

SECONDARY OUTCOMES:
Diagnostic accuracy of T1-,T2- and diffusion-mappings deriving from MRF in myometrial invasion detection | 3 months
Correlation between T1-, T2- and diffusion mappings and DFS and OS | 3 years
Diagnostic accuracy of T1-,T2- and diffusion-mappings and pathological nodal involvement | 3 months
Evaluation of Radiomic and Radiogenomic models to predict recurrence in early stage EC and to predict DFS and OS | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Universitaro "A. Gemelli" IRCCS, Roma, Italy